CLINICAL TRIAL: NCT00714805
Title: Non-Invasive Measurement of GI Motility in Patients With ALS
Brief Title: Non-Invasive Measurement of Gastrointestinal (GI) Motility in Patients With Amyotrophic Lateral Sclerosis (ALS)
Acronym: GIDysmotility
Status: Completed | Type: Observational
Sponsor: Christine Barr (Other)
Collaborators: MDA/ALS Center of Hope (Other)
Responsible Party: Sponsor-Investigator, Christine Barr, Primary contact, Drexel University
Organization: Drexel University (Other)
Other Study IDs: Internal-16637
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Gastric Motility; Autonomic Nervous System; Neurodegenerative Diseases; Movement Disorders; Gastrointestinal Motility
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases; Movement Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ALS: Subjects having either definite or probable ALS by El Escorial Criteria.
- Healthy Control: Subjects having no known ailment.

SUMMARY:
Recent evidence implicates abnormalities of autonomic function in ALS including problems with gastrointestinal (GI) motility. GI complaints reported by ALS patients such as constipation, diffuse abdominal pain, and a feeling of fullness or nausea may be attributed to autonomic involvement. Toepfer et al. found delayed gastric emptying in most ALS patients, indicating autonomic dysfunction (Gastrointestinal dysfunction in amyotrophic lateral sclerosis. Amyotrophic Lateral Sclerosis Other Motor Neuron Disord 1999; 1:15-19). The same authors also reported markedly prolonged colon transit time in ALS (Toepfer et al: Delayed colonic transit times in amyotrophic lateral sclerosis assessed with radio-opaque markers. Eur J Med Res 1997; 2:473-476).

The present study will investigate the GI transit time in a large cohort of patients and controls using a noninvasive technique that measure hydrogen gas production with the digestion of lactulose in a measured substrate load presented to the bowel.

DETAILED DESCRIPTION:
This study will examine how much time it takes for the food to travel along the intestines from mouth or stomach (if you have a feeding tube) to the end of the large intestine using a special instrument that measures hydrogen gas in your breath. Data collection will start after you sign this consent form. The only procedures that would be above and beyond routine care are indicated below:

In order to prepare for the study you will be asked to be off all medications that affects the GI motility for 24 hours. You will also be asked to fast overnight (starting midnight) the day before the test.

After fasting overnight, the test will be performed in the morning (at the Neurology Outpatient Clinic or at your home). Before eating or drinking anything a baseline measurement will be taken by breathing into the hydrogen meter. This will be just normal breathing. You will then drink a test meal consisting of 250 ml (approximately 1 cup) of a lactose (type of sugar) free supplement (For example Ensure) that has 20 grams of Lactulose added. If you have a peg tube then the supplement will be given through the tube. After 10 minutes you will again be asked to breath into the machine to measure the hydrogen gas levels. This will be repeated every 10 minutes until the hydrogen levels rise to a certain level or until 4 hours have passed.

ELIGIBILITY:
Inclusion Criteria:

For the Disease Population:

* Diagnosis of definite or possible ALS by the El Escorial Criteria
* No previously known gastrointestinal problems
* Able to fast and hold medicines (anticholinergics and prokinetics) overnight prior to the measurement of GI motility
* No unstable medical problems and no evidence of dehydration by examination (skin turgor)

For Healthy Control

* No known gastrointestinal illness
* Able to fast and hold medicines (anticholinergics) overnight prior to the measurement of GI motility
* No unstable medical problems or evidence of dehydration

Exclusion Criteria:

* Patients or controls who are dehydrated
* Patients or controls who have evidence of previous gastrointestinal disease
* Patients with any unstable medical condition
* Patients unable to give informed consent
* Patients unable to blow into the breath analyzer and have steady breathing for one minute

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ALS clinic patients at MDA/ALS Center of Hope.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2007-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
GI Transit Time | 1 session
  GI Transit Time is determined by measuring the levels of hydrogen gas in exhaled breath using a Hydrogen Meter.

CONTACTS AND LOCATIONS:
Overall Officials: Terry D Heiman-Patterson, MD, Principal Investigator — Drexel University College of Medicine
Locations (1):
- MDA/ALS Center of Hope, Philadelphia, Pennsylvania, United States